CLINICAL TRIAL: NCT00901043
Title: Effects of Walnut Consumption on Endothelial Function in Type 2 Diabetes: A Randomized, Controlled, Cross-over Trial
Brief Title: Effects of Walnut Consumption on Endothelial Function in Type 2 Diabetes
Acronym: WALNUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2007-10
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: DIABETES MELLITUS TYPE 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walnut supplementation (Experimental): Eight weeks with walnut supplementation to an ad lib diet
  Interventions: Dietary Supplement: Walnut supplementation
- Ad lib diet (Active Comparator): Eight weeks ad lib diet without walnut supplementation
  Interventions: Dietary Supplement: Ad lib diet

INTERVENTIONS:
Dietary Supplement: Walnut supplementation — Eight weeks of walnut supplementation
  Arms: Walnut supplementation
Dietary Supplement: Ad lib diet — Eight weeks without walnut supplementation
  Arms: Ad lib diet

SUMMARY:
The purpose of this study is to examine the effects of sustained walnut consumption on endothelial function and lipid markers in patients with Type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Evidence-based guidelines for the management of type 2 diabetes mellitus and related cardiovascular disease (CVD) refer to cardioprotective dietary fatty acid proportions. Several studies demonstrate the hypocholesteremic effects of walnuts in energy restricted diets. To our knowledge, the health benefits accrued as a result of addition of walnuts to an ad libitum diet in type 2 diabetic subjects have not been studied. Addition of walnuts to an ad libitum diet represents a practical way to achieve the recommended fatty acid proportions. The proposed study will examine whether a total dietary pattern inclusive of walnuts, will result in amelioration of cardiac risk as measured by improvement in endothelial function and glycemic control in type 2 diabetics. Results of the study will have important implications for clinicians and dietitians in dietary management of type 2 diabetes. Demonstrating that walnuts can be regarded as beneficial components of dietary management of type 2 diabetes is of relevance to the walnut industry as well. The study employs a pragmatic approach to approximate dietary practices in a real world setting thus enhancing the external validity of the study. If positive, the study results can inform future marketing efforts of the California Walnut Commission. Demonstrating that addition of walnuts to an ad libitum diet can potentially lead to improvement in endothelial function, improve lipid profiles, glycemic control and reduce the risk of CVD complications in diabetic patients has important applications for dietary management of diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. men and women ages 35-75
2. non-smoker
3. able to have blood pressure taken bilaterally
4. diagnosed with type 2 diabetes by physician for at least one year
5. stable glucose levels and medication dose for the past 3 months
6. not on insulin therapy

Exclusion Criteria:

1. failure to meet inclusion criteria
2. anticipated inability to complete or comply with study protocol for any reason (e.g., inability to communicate in English, dementia) or any unstable medical condition that would limit the ability of a subject to participate fully in the trial (e.g., wasting illness, AIDS, tuberculosis, psychotic disorder)
3. diagnosed eating disorder
4. use of lipid-lowering or antihypertensive medications (statins, red rice yeast extract, garlic) unless stable on medication for at least 3 months and willing to refrain from taking medication for 12 hours prior to endothelial function (EF) scanning, vasoactive medication (i.e., glucocorticoids, antineoplastic agents, psychoactive agents, or bronchodilators) or nutriceuticals
5. regular use of multivitamins and/or complementary or alternative supplement therapy and unwillingness to discontinue supplementation for at least 8 weeks prior to study initiation and for study duration
6. any rheumatologic disease requiring regular use of nonsteroidal antiinflammatory drug (NSAIDs) or alternative medications
7. regular use of fiber supplements
8. preexisting cardiovascular disease, including symptomatic coronary artery disease (CAD), myocardial infarction, angina pectoris, anginal equivalent, peripheral vascular disease (claudication, amputation, or revascularization) congestive heart failure, carotid stenosis, aortic stenosis or stroke; diabetes, sleep apnea, severe uncontrolled hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 105 mmHg)
9. coagulopathy, known bleeding diathesis or history of clinically significant hemorrhage; current use of warfarin
10. clinically significant anemia (Hct < 36% in men, < 33% in women)
11. intestinal or stomach disease
12. inability to use right or left arm for endothelial function testing for any reason such as breast surgery, trauma, radiation to right axilla, lymphedema, right arm shunt, severe vascular disease in right arm
13. subjects on a disease specific diet
14. subjects on a weight control diet
15. subjects on a vegan diet
16. allergy to any kind of nut, including walnuts and peanuts

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow mediated dilation (FMD) | 8 weeks

SECONDARY OUTCOMES:
Change in weight, waist circumference, blood pressure, fasting lipids, fasting insulin, HBA1c and glucose levels | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: DAVID L KATZ, MD, Principal Investigator — Yale-Griffin Prevention Research Center
Locations (1):
- Griffin Hospital, Derby, Connecticut, United States